CLINICAL TRIAL: NCT00042172
Title: Cognitive Enhancers Explored With PET Imaging
Brief Title: Treatment for Early Memory Loss
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21MH061801 (NIH); R21MH061801 (NIH); DSIR AT-GP
Record Dates: First submitted 2002-07-24; First posted 2002-07-26 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Cognition Disorders; Alzheimer Disease
Keywords: Cognition; Memory
MeSH Terms: conditions — Cognition Disorders; Alzheimer Disease | interventions — Donepezil; Ginkgo biloba extract

INTERVENTIONS:
Drug: Donepezil
Drug: Ginkgo Biloba Extract

SUMMARY:
The purpose of this study is to evaluate the effectiveness of donepezil (Aricept) for the treatment of mild cognitive impairment (MCI) in elderly adults. This study will also determine whether adding ginkgo biloba extract (GBE) enhances the effects of donepezil.

DETAILED DESCRIPTION:
Cognition involves important thinking processes such as perception, learning, and reasoning. There are currently no definitive treatments for cognitive deterioration. This study focuses on elderly individuals with MCI because people at a pre-dementia stage may sustain the greatest and most lasting benefit from cognitive-enhancing agents.

Patients receive either donepezil or placebo for the first 6 months of the study. In the second 6 months of the study, patients are randomized to receive either donepezil plus GBE or donepezil alone. Positron Emission Tomography (PET), which provides a color-coded image of the brain's blood flow in a particular area, is used to assess brain activity during memory tasks. A PET scan is performed at study entry, 6 months, and 1 year. A vasodilator (a drug that dilates the blood vessels) is administered during the PET imaging procedure to determine whether vascular disease affects memory function. A magnetic resonance imaging (MRI) scan is also taken to view the brain.

ELIGIBILITY:
Inclusion Criteria:

* Display impairment on at least 2 of 3 memory tests
* Meet the following criteria for mild cognitive impairment: subjective complaint of memory problems; no impairment in activities of daily living; general cognitive function in the normal age-adjusted range; abnormal memory function for age; and lacking full DSM criteria for dementia

Exclusion Criteria:

* Have a history of major neurological, metabolic, psychiatric or cardiovascular disease (patients with a history of non-CNS oncologic disease treated surgically and currently in remission will not be excluded)
* Have a cerebrovascular condition
* Abuse alcohol or drugs
* Have renal or hepatic disease, diabetes mellitus, gout, or adrenocortical insufficiency
* Are sensitive to carbonic anhydrase inhibitors, antibacterial sulfonamides, thiazide diuretics, or other sulfonamide-derivative diuretics
* Have taken donepezil or GBE products prior to enrollment
* Have taken medications, including herbal agents (exceptions will be made for routine health maintenance medications such as alendronate [Fosamax] for osteoporosis, vitamin therapy [not to exceed 200 percent RDA for any particular vitamin], thyroid replacement therapy, hormone replacement, and ophthalmic medications for glaucoma and other eye disorders)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40
Dates: Start 2002-06; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Department of Psychiatry, Iowa City, Iowa, United States